CLINICAL TRIAL: NCT04846699
Title: Triangulation, Eye of the Needle and Stone Direct Targeting Percutaneous Renal Access Techniques of Nephrolithotomy : Randomized Controlled Trial
Brief Title: Triangulation Bulls Eye and Stone Direct Targeting Pcnl
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mahmoud eldardery, dr mahmoud abdo el dardery, Assiut University
Other Study IDs: new pcnl approch
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Endourology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: bulls eye localization
  Interventions: Procedure: per-cutaneous stone extraction
- group 2: stone targeted technique renal access
  Interventions: Procedure: per-cutaneous stone extraction
- group 3: triangulation renal access technique
  Interventions: Procedure: per-cutaneous stone extraction

INTERVENTIONS:
Procedure: per-cutaneous stone extraction — percutaneous nephrolithotripsy for renal stones by different renal access

SUMMARY:
To assess the impact of percutaneous renal access technique on outcomes of percutaneous nephrolithotomy in management of renal stones by comparing the Triangulation and ''eye of the needle'' (or bull's eye) and the stone targeted techniques in the following:-

1. Stone free rate (SFR) (primary outcome).
2. Complicatins of surgery (primary outcome).
3. Change in haematocrit pre and postoperative (secondary outcome).
4. Operative time (secondary outcome).
5. Duration of hospitalization (secondary outcome). .

7-Fluroscpic screening time (FST) (secondary outcome). . 8- Change in haematocrit pre and postoperative (secondary outcome).

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PNL) is an appropriate first-line alternative for the management of kidney stones that are larger than 2 cm in diameter and that do not respond to extracorporeal shock wave lithotripsy (SWL) [1,2].

Percutaneous renal access is the most important step in PNL, and the adequacy of access directly affects the success and complication rates of this procedure.

Among C-arm fluoroscopy, computed tomography (CT), and ultrasonography (US), C-arm fluoroscopy is the most commonly used imaging technique to access the intrarenal collecting system [3-4].

Various fluoroscopy techniques have been described for achieving a good access. One can use fluoroscopy or ultrasonography or a combination of both for reaching the target calyx. Each of it has its advantages and disadvantages, and no consensus exists showing the superiority of one or the other [5].

Triangulation and ''eye of the needle'' (or bull's eye) techniques are two common methods to obtain proper percutaneous renal access under fluoroscopy guidance [6-7].

Multiplanar fluoroscopic imaging is essential in both techniques to make a proper renal puncture.

Biplanar access is based on mediolateral and cephalad-caudal movements of the needle, with the depth of the puncture adjusted based on different fluoroscopic projections, including oblique, vertical, and 30° positions [6, 8].

Most published studies of PCNL have focused on evaluating the effect of patient- and stone-related factors such as success rate, extent of bleeding, complication rate, fluoroscopic Screening times (FSTs), and operative time on outcomes. [9-10]

The imaging modalities used for guidance by urologists or radiologists during percutaneous renal access and renal access procedures have also recently been analyzed and compared in terms of outcomes and complications.[11-12]

These studies, however, have not considered the effect of percutaneous renal access technique on outcome. Although the triangulation and the bull's-eye techniques have been evaluated and compared using a biologic model in a published study [13], no clinical study comparing these techniques has been performed.

The aim of this study is to evaluate the impact of percutaneous renal access technique on outcomes of percutaneous nephrolithotomy in management of renal stones by comparing the Triangulation and ''eye of the needle'' (or bull's eye) and the stone targeted technique .

ELIGIBILITY:
Inclusion Criteria:

- The study will include all adult patients that with renal stones larger than 2 cm in diameter who will attend our endourology outpatient clinic from Jan 2021 to February 2023 and consented to participate in the study.

Exclusion Criteria:

- 1-Patients with urinary system anomalies as horseshoe kidney, ectopic pelvic kid.

2-Patients with skeletal malformations. 3-Bleeding tendency and ongoing anticoagulant therapy. 4-Pregnancy. 5-Patients who refuse to be involved in the trial documentation.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: all patients presented to endourology clinic by renal stone and complianting and fit for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
stone free rate | 48 hours postoperative
  outcome of residual stone postoperative
complication of surgery | from day one post-operative to 3 months
  fever , urine leakage , stent of ureter , sepsis, other intervention

CONTACTS AND LOCATIONS:
Locations (1):
- NIH, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmahl FW, Betz E, Talke H, Hohorst HJ. [Energy rich phosphates and metabolites of energy metabolism in the cerebral cortex in the cat]. Biochem Z. 1965 Sep 30;342(5):518-31. No abstract available. German. PMID 5866850
- [Background] Ashley FL. Implications of wound healing research. A meeting ground for experimental biology and clinical medicine. Plast Reconstr Surg. 1969 Feb;43(2):190-1. No abstract available. PMID 5765923
- [Background] Meshkov SL, Seltzer SE, Finberg HJ. CT detection of intraabdominal disease in patients with lower extremity signs and symptoms. J Comput Assist Tomogr. 1982 Jun;6(3):497-501. doi: 10.1097/00004728-198206000-00010. PMID 7096695